CLINICAL TRIAL: NCT05767671
Title: Macrophage Programing in Acute Lung Injury
Brief Title: Macrophage Programing in Acute Lung Injury: MiniBAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Janssen, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, William Janssen, MD, Section Head of Critical Care, Professor of Medicine, Principle Investigator, National Jewish Health
Organization: National Jewish Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS3076
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilator Associated Pneumonia
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: The population to be studied are patients identified to have ARDS, admitted to the intensive care unit, and placed on a mechanical ventilator. Control subjects will be individuals on mechanical ventilation for non-pulmonary reasons (i.e. following surgery, sepsis without lung involvement). A total of 56 subjects will be enrolled. As described below (in Research Methods and Enrollment) a 2:1 ratio of ARDS to control subjects will be targeted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population Group (Other): People in the ICU on mechanical ventilation due to a diagnosis of ARDS or any other diagnosis that requires mechanical ventilation (following surgery, sepsis without lung involvement, seizures)
  Interventions: Other: Non-Bronchoscopic Mini Bronchoalveolar Lavage

INTERVENTIONS:
Other: Non-Bronchoscopic Mini Bronchoalveolar Lavage — A minimally invasive technique frequently used in the ICU to obtain alveolar fluid samples from mechanically ventilated patients. The technique uses a commercially available telescoping catheter with a curved distal tip that allows the operator to direct the catheter into the right or left lung. The catheter is passed through an air-tight adapter on the distal end of the endotracheal tube and gently advanced to the desired lung until resistance is encountered. The inner catheter is then advanced until resistance is again encountered, signifying that the distal catheter tip is "wedged." 20ml of sterile saline is instilled into the catheter followed by 5 ml of air, and the fluid aspirated. Two additional 20ml aliquots of sterile saline are injected and aspirated in a similar fashion. Specimens are pooled and on average provide a combined volume of 10ml.

SUMMARY:
The goal of this observational clinical trial is to learn about the role white blood cells (macrophages) play in lung inflammation in people with Acute Respiratory Distress Syndrome (ARDS). The main questions it aims to answer are:

1. How does the immune system respond to different kinds of lung injury and inflammation and how do those processes differ from each other?
2. What roles do the cells that live in the lungs (macrophages) play in turning off inflammation? How does their role differ from other cells that are called to the lung to help repair injury (recruited macrophages)?
3. Will more frequent testing of lung cell samples help reduce the time it takes to start treatment for ventilator-associated pneumonia (VAP) and therefore reduce the rates of initial therapy failure?

Participants will be in the intensive care unit (ICU) on a mechanical ventilator (machine that helps patients breathe) because they have ARDS or are on a mechanical ventilator for some other reason (control group). The following will happen:

1. Participants will be given 100% oxygen through the breathing machine (mechanical ventilator) for 3-5 minutes. This is called pre-oxygenation.
2. A lung specialist (pulmonologist), a member of Dr. Janssen's research team, or respiratory therapist will place small amount of saline into the lung using a long catheter going through the breathing tube.
3. The fluid will be removed with suction and will be sent to the laboratory for testing.
4. This will be repeated two more times over the course of 10 days, or less if participants are taken off of the ventilator. The procedure will be performed no more than three times.
5. Two nasal brushings will be taken from the participants' nose.
6. Approximately 3 tablespoons of blood will be removed by putting a needle into the participants vein. This is the standard method used to obtain blood for tests. A total of 9 tablespoons will be taken for research purposes over the course of this study
7. Data including the participants age, sex, severity of illness, and other medical conditions will be recorded to determine how these can affect the white blood cells.
8. If bacteria are isolated from the fluid in the participants lung, the participants' physician may choose to place the participants on antibiotics to treat an infection.
9. A follow-up phone call may be made by a member of the research team after discharge from the hospital. At this time, the participant may be invited to participate in the Post-ICU clinic at National Jewish Health.

DETAILED DESCRIPTION:
This research study is looking at the role of white blood cells in acute respiratory distress syndrome (ARDS). ARDS is a severe, life-threatening disease caused by uncontrolled inflammation in the lungs. Macrophages are a type of white blood cell that is involved in both causing and removing inflammation. The goal of this study is to learn more about macrophages in the setting of ARDS, so that the investigators can potentially find new treatments for this disease. To get the best information for this study, macrophages from patients with ARDS will be compared to macrophages from individuals with healthy lungs.

All participants in this study must be on a breathing machine (mechanical ventilator). Participants must either have damage to the lungs (ARDS) or have healthy lungs with no prior history of lung disease. Participants must fit into one of these categories. For this study, the investigators will isolate macrophages from a sample of fluid obtained from the lungs. While the method used to obtain the sample of fluid is a standard procedure performed in the ICU, the investigators will be performing it for research purposes. The investigators will also be collecting two nasal brushes. During the nasal brushing a small brush will be inserted into the first one or two inches of the participants nasal cavity from the participants nostril by a member of the research team. The brush will be moved back and forth gently, then removed. A second brush will be inserted in the other nostril and the technique repeated. A second part of our study is to determine whether regularly sampling fluid from the lungs and looking for bacteria will help us catch and treat pneumonia quicker. As such, a portion of the fluid obtained from the lungs, will be sent to the laboratory to look for bacteria growing in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (by LAR if subject unconscious or has altered mental status) prior to any study procedures. Verbal consent may be used as necessary
* Adults greater than 18 years of age
* Admission to the intensive care unit.
* Orally/nasally intubated or expected to be intubated within 48 hours

Exclusion Criteria:

* History of solid organ or bone marrow transplantation
* Severe or massive hemoptysis
* At significant risk for bleeding (INR > 3 or PTT > 3x normal)
* Presence of pneumomediastinum or pneumothorax on recent imaging
* Presence of an advanced directive with Do Not Intubate (DNI) status (Do Not Resuscitate (DNR) is acceptable)
* Morbid state or expected to survive less than 24 hours because of an advanced co-morbid medical condition in the opinion of the PI and/or clinical team and attending physician.
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate host response to ARDS | Days on ventilator 1-2, 4-6 and 8-10
  Compare host response due to ARDS caused by COVID19 versus other forms of ARDS and to determine how resident and recruited macrophages influence inflammation during ARDS and how they differentially contribute to lung repair.
Macrophage signaling | Days on ventilator 1-2, 4-6 and 8-10
  1. The host response to COVID19 includes a robust inflammatory response with exceedingly high levels of pro-inflammatory cytokines such as IL-6. We hypothesize that macrophage signaling plays a major role in these responses.
Resident alveolar Macrophages | Days on ventilator 1-2, 4-6 and 8-10
  2. Resident alveolar macrophages will remain constant in number throughout the course of ARDS whereas recruited macrophages will increase in number and then ultimately undergo apoptosis as inflammation resolves. Alveolar macrophages will be isolated from mini BAL of ARDS subjects and mechanically ventilated controls. Macrophage subsets will be distinguished with flow cytometry and enumerated.
Recruited versus resident macrophages | Days on ventilator 1-2, 4-6 and 8-10
  3. Recruited macrophages from ARDS subjects will be more pro-inflammatory than resident macrophages at early time points (i.e. days 1-2) and produce pro-reparative molecules at later time points. Macrophage subsets will be isolated using FACS and subjected to RNA sequencing. Pro-inflammatory and pro-reparative modules will be assessed in the data set expression of transcription factors reported to drive macrophage polarization (HIF-1α, NF-kB, STAT-1, STAT-3, STAT-6, PPARγ, PU.1) will be assessed. Macrophages from control subjects will be used to determine baseline activation and transcriptional status.

SECONDARY OUTCOMES:
Ventilator associated pneumonia (VAP) | Days on ventilator 1-2, 4-6 and 8-10
  A secondary objective of the study is to reduce time to diagnosis and treatment of ventilator-associated pneumonia (VAP) in an at risk population. All patients on mechanical ventilation are at risk for developing VAP. Prompt administration of antibiotics has been shown to improve mortality. Accordingly appropriate selection of anti-microbial agents is paramount. To assess potential microbial pathogens in the lungs, a 1ml aliquot of each mini-BAL will be sent to the microbiology lab at National Jewish - St. Joseph Hospital to obtain quantitative bacterial cultures, bacterial speciation, and antibiotic sensitivity profiles. These results will be made available to the treating physician and can be used to aid in antibiotic selection and administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Health - St. Joseph's Hospital - National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No